CLINICAL TRIAL: NCT00493896
Title: Safety of Fondaparinux as Routine VTE Prophylaxis in Medical ICU Patients: An Investigator Initiated Protocol
Brief Title: Safety of Fondaparinux as Routine VTE Prophylaxis in Medical ICU Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 107696
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism Prophylaxis; VTE prophylaxis
MeSH Terms: conditions — Venous Thromboembolism | interventions — Fondaparinux; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fondaparinux (Experimental): Fondaparinux treatment - one standard of care option
  Interventions: Drug: Fondaparinux
- 2 (Active Comparator): Enoxaparin
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Fondaparinux — The dose for Arixtra is 2.5 mg once daily, subcutaneously.
  Other Names: Arixtra
  Arms: Fondaparinux
Drug: Enoxaparin — The dose for Lovenox is 40 mg once daily, subcutaneously.
  Other Names: Lovenox
  Arms: 2

SUMMARY:
This is a pilot study to evaluate safety of fondaparinux and enoxaparin in terms of bleeding and development of thrombocytopenia in the medical ICU population.

DETAILED DESCRIPTION:
This is a pilot study to evaluate safety of fondaparinux and enoxaparin in terms of bleeding and development of thrombocytopenia in the medical ICU population. We expect the null hypothesis to be proven true. One hundred subjects will be enrolled in this prospective, randomized, double-blind (concealed allocation) pilot study of consecutive medical ICU patients to one of two pharmacologic VTE prophylaxix treatment arms. (1) Primary endpoints include hemoglobin, hematocrit, & platelet counts. blood product utilization, bleeding complications (any), Steady State Functional Factor Xa activity (for post hoc analysis), non-study pharmacologic VTE prophylaxis (when estimated CLcr < 30ml/min), and days not treated with study drug or treated with alternative agent Secondary/ Additional Data to be collected include patient demographics, primary & secondary diagnoses, central venous access, and sequential compression device utilization.

ELIGIBILITY:
Inclusion Criteria:

1. Ability or legally authorized representative (LAR) to provide informed consent
2. Adult who has not had surgery within 10 days, admitted to the Sentara Norfolk General Hospital ICU Medical Teaching Services for any reason.

Exclusion Criteria:

1. Active or suspected bleeding
2. Platelet count less than 100,000 per microliter (mm3) of blood
3. Thrombolytic or anticoagulant treatment (including any doses of prophylactic UFH, LMWH or fondaparinux) during the current hospitalization
4. Initial estimated CLcr < 30 ml/min as determined by the Cockcroft-Gault equation
5. Initial labs indicative or suggestive of rapidly rising serum Creatinine (>1 mg/dL/day)
6. Pregnancy (for medicolegal considerations)
7. Patients with or expecting to require an epidural catheter
8. Patients who are expected to have an immediate (within 24h) need for surgery

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Bleeding events | inpatient hospitalization

SECONDARY OUTCOMES:
Development of thrombocytopenia | inpatient hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Callender, MD, Principal Investigator — Eastern VA Medical School, Norfolk, VA